CLINICAL TRIAL: NCT05570214
Title: Impact of Virtual Reality on Patient Vital Signs During Urological Bedside Vasectomies
Brief Title: A Study of Virtual Reality During Urological Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of PI interest
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David D. Thiel, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-000947
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Virtual Reality; Vasectomy Procedure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Group (Experimental): Subjects will wear a virtual reality headset during their urological bedside vasectomy.
  Interventions: Other: Virtual Reality
- Standard of Care Group (No Intervention): Subjects will undergo standard of care urological bedside vasectomy

INTERVENTIONS:
Other: Virtual Reality — Virtual reality device will be viewing calming narrated scenarios with relaxing music of walking through a forest, along a beach, through a Chinese garden, a winter landscape or taking off in a spaceship or snorkeling through a reef
  Arms: Virtual Reality Group

SUMMARY:
This research is being done to see if virtual reality devices are able to distract patients during Urologic beside vasectomy procedures in the clinic and help improve patient experience and vital signs.

DETAILED DESCRIPTION:
Once participants are consented and checked in for the procedure, researchers will obtain the randomization assignment from a REDCap database with a randomization module designed by the study statistician. Participants will be randomized in a 1:1 ratio to either virtual reality or standard of care.

Researchers will collect participant vital signs (heart rate, blood pressure, and SpO2) at check in, laying down on the table, in the midst of the procedure, and after the procedure is complete. After the procedure is completed, all participants will be given two surveys about satisfaction with the experience to complete. Researchers will record any medications the participants takes the day of the procedure. Researchers will then gather demographic data from the participant's chart through Epic (age, height, weight, BMI, race, ethnicity, past medical history, and procedure information). All study data will be stored in a secure REDcap database. Researchers have teamed up with members of the anesthesia department at Mayo Clinic Florida who have performed similar studies utilizing the virtual reality headsets. The department has three virtual reality headsets and know how to operate them.

The participants who are selected to use the virtual reality device will be viewing calming narrated scenarios with relaxing music of walking through a forest, along a beach, through a chinese garden, a winter landscape or taking off in a spaceship or snorkeling through a reef.

ELIGIBILITY:
Inclusion Criteria:

- Any patient undergoing a vasectomy, transrectal prostate biopsy, cystoscopy, Doppler ultrasound, or Xiaflex.

Exclusion Criteria:

- Anyone < 18 years of age.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | Baseline, intra-procedure, post-procedure (approximately 1 hour)
  Number of beats per minute
Change in Systolic blood pressure | Baseline, intra-procedure, post-procedure (approximately 1 hour)
  Measured in millimeters of mercury (mmHg)
Change in diastolic blood pressure | Baseline, intra-procedure, post-procedure (approximately 1 hour)
  Measured in millimeters of mercury (mmHg)
Change in oxygen saturation levels | Baseline, intra-procedure, post-procedure (approximately 1 hour)
  Measured by a pulse oximeter reading reported as a percentage

SECONDARY OUTCOMES:
Patient satisfaction | Post-procedure (approximately 1 hour)
  Measured using the self-reported QoR-15 patient survey. 15-item questionnaire used to assess feelings and pain within the last 24 hours on a scale from 0 to 10; 0 indicating none of the time [poor] and 10 indicating all of the time [excellent]. Higher total scores indicate greater patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: David Thiel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials